CLINICAL TRIAL: NCT07390929
Title: Clinical Trial Study on the Improved New Method of Acupotomy for Ankylosing Spondylitis
Brief Title: Clinical Trial Study on the Improved New Method of Acupotomy for AS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henan Provincial People's Hospital (Other)
Collaborators: The Second Affiliated Hospital of Henan University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, zhouzipeng, Chief physician, The Second Affiliated Hospital of Henan University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025YFC3508501
Record Dates: First submitted 2026-01-29; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-07

CONDITIONS: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): All subjects were enrolled at week 0 and, after completing baseline assessments, received acupotomy treatment once per week for a total of four sessions over the initial three-week period. The core intervention for the treatment group (acupotomy group) involved ultrasound-guided precise release: first, the target vertebra with the most significant lesions was identified through palpation and ultrasound imaging, after which the acupotomy was accurately guided in real-time via ultrasound to the interspinous points (located at the interspinous ligaments) and paraspinal points (located at the intertransverse ligaments) of the target vertebra and adjacent vertebrae for release.
  Interventions: Procedure: Acupotomy
- Control Group (Sham Comparator): The control group (sham acupotomy group) strictly replicated all preliminary procedures of the treatment group, including exploration, ultrasound localization, and local anesthesia. However, the acupotomy needle only pierced the epidermis without performing any release operations in the deeper tissues, thereby maintaining blinding and assessing the specific effect of the acupotomy therapy.
  Interventions: Procedure: Sham Acupotomy

INTERVENTIONS:
Procedure: Acupotomy — All subjects were enrolled at week 0 and, after completing baseline assessments, received acupotomy treatment once per week for a total of four sessions over the initial three- week period. The core intervention for the treatment group (acupotomy group) involved ultrasound-guided precise release: first, the target vertebra with the most significant lesions was identified through palpation and ultrasound imaging, after which the acupotomy was accurately guided in real-time via ultrasound to the interspinous points (located at the interspinous ligaments) and paraspinal points (located at the intertransverse ligaments) of the target vertebra and adjacent vertebrae for release.
  Arms: Treatment Group
Procedure: Sham Acupotomy — The control group (sham acupotomy group) strictly replicated all preliminary procedures of the treatment group, including exploration, ultrasound localization, and local anesthesia. However, the acupotomy needle only pierced the epidermis without performing any release operations in the deeper tissues, thereby maintaining blinding and assessing the specific effect of the acupotomy therapy.
  Arms: Control Group

SUMMARY:
This study employs a randomized controlled trial methodology to systematically evaluate the efficacy and safety of a modified acupotomy technique in the treatment of ankylosing spondylitis. Through ultrasound-guided localization, the operative sites are assessed to clarify the improvement effect of the modified acupotomy on disease activity in AS patients. The aim is to enhance the clinical outcomes of AS, provide evidence-based medical support for acupotomy treatment of AS, and improve the diagnosis and treatment standards for the condition.

ELIGIBILITY:
Inclusion Criteria:

1. Meeting the revised New York Criteria (1984) or the Assessment of SpondyloArthritis international Society (ASAS) classification criteria for axial spondyloarthritis (2009).
2. Aged 18 to 75 years old.
3. Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) score ≥ 4 points.
4. Having signed the informed consent form.

Exclusion Criteria:

1. Complicated with other autoimmune diseases except for the research disease.
2. Complete ankylosis or deformity of the spine.
3. Pregnant or lactating women.
4. Complicated with severe cardiovascular and cerebrovascular diseases, liver or kidney failure, malignant tumors, or coagulation disorders.
5. Patients whose data collection is affected by mental, language or other factors.
6. Patients with psoriatic arthritis, reactive arthritis, or inflammatory bowel disease-associated spondyloarthritis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11-05 (Actual); Primary Completion 2028-07-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Bath Ankylosing Spondylitis Disease Activity Index | Week 0, Week 2, Week 4, Week 8
  Based on the patient's symptoms over the past week, an assessment is conducted through six questions. The first five questions are scored using a Visual Analog Scale (VAS, 0-10 points). The calculation formula is generally expressed as: BASDAl = 0.2x(A+B+C+D+(E+ F)/2) Where: A represents the degree of fatigue/tiredness; B represents the degree of pain in the neck, back, or hips; C represents the degree of pain/swelling in other joints; D represents the level of discomfort from bodily tenderness or pressure pain; E represents the severity of morning stiffness; F represents the duration of morning stiffness (converted to a 0-10 score). BASDAI 24 indicates high disease activity, while a score <4 suggests lower disease activity.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Henan University of Chinese Medicine, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No